CLINICAL TRIAL: NCT01487031
Title: Assessment of the Use of Music Therapy on Nausea and Pain During Hospitalization for Autologous Stem Cell Transplantation
Brief Title: Music Therapy on Nausea and Pain for Autologous Stem Cell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CASE11Z10
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Multiple Myeloma; Non-Hodgkin Lymphoma; Hodgkin Lymphoma
Keywords: Autologous Stem Cell Transplantation; multiple myeloma; non-Hodgkin; Hodgkin lymphoma; Music Therapy; Nausea; Pain
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Nausea; Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music Therapy (Experimental): Patients randomized to receive music therapy will receive 2 sessions of live music therapy, at least 48 hours apart, from a Music Therapist-Board Certified (MT-BC, certified through the Certification Board for Music Therapists) in their room.
  Interventions: Other: Music Therapy
- No music therapy (Active Comparator): Those patients randomized to standard therapy (no music therapy) are allowed to listen to music; however they will not receive interactive music therapy from a certified therapist.
  Interventions: Other: No music therapy

INTERVENTIONS:
Other: Music Therapy — Patients randomized to receive music therapy will receive 2 sessions of live music therapy, at least 48 hours apart, from a Music Therapist-Board Certified (MT-BC, certified through the Certification Board for Music Therapists) in their room
  Arms: Music Therapy
Other: No music therapy — Those patients randomized to standard therapy (no music therapy) are allowed to listen to music; however they will not receive interactive music therapy from a certified therapist.
  Arms: No music therapy

SUMMARY:
Autologous stem cell transplant (ASCT) is an important therapy for patients with multiple myeloma, non-Hodgkin's lymphoma, and Hodgkin's lymphoma. It has been shown to improve progression free survival and overall survival. However, it is a challenging treatment process both physically and psychologically. It is a procedure with many side effects that can be uncomfortable, painful, and at times, difficult to endure. Complementary therapies, such as music therapy, have potential to be an important adjunct in palliation of symptoms in patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Patients randomized to receive music therapy will receive 2 sessions of live music therapy, at least 48 hours apart, from a Music Therapist-Board Certified (MT-BC, certified through the Certification Board for Music Therapists) in their room. This will occur between days -1 and +5, with the first music therapy session being as close to day +1 as possible and the second session being at least 48 hours later (but no more than 96 hours later).

Those patients randomized to standard therapy (no music therapy) are allowed to listen to music; however they will not receive interactive music therapy from a certified therapist. Following day +7, music therapy will be offered to all patients who are interested in participating.

No narcotic or anti-emetic therapy will be administered for at least 2 hours prior to music therapy sessions or to assessments. Patients will rate nausea and pain at the beginning and end of the first music therapy session on a validated visual analog scale.12-14 The scale will be 10cm with the least nausea or pain at point 0 and the greatest nausea or pain at point 10. Patients will be asked to rate their nausea and pain on day +5 and day +7.

ELIGIBILITY:
Inclusion Criteria:

* Be older than 18 years of age
* Have a diagnosis of multiple myeloma, non-Hodgkin, or Hodgkin lymphoma
* Be undergoing ASCT (Autologous Stem Cell Transplantation)

Exclusion Criteria:

* Have had previous ASCT
* Have a diagnosis of leukemia
* History of prior music therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Patient perception of nausea | 7 days after intervention
  Compare the difference in patient perception of nausea in those who receive music therapy and those who do not.
Patient perception of pain | 7 days
  Compare the difference in patient perception of pain in those who receive music therapy and those who do not.

SECONDARY OUTCOMES:
Quality of life | 7 days
  Compare mood disturbance and quality of life in those who receive music therapy and those who do not.
Use of "as needed" narcotic medications | 7 days
  Compare the difference in the use of "as needed" narcotic medications in those who receive music therapy and those who do not (using morphine equivalent doses).
Monitoring of physiologic responsiveness | 7 days
  Compare non-invasive monitoring of physiologic responsiveness to provide an index of autonomic nervous system function, or general arousal. We hypothesize that arousal will decrease after music therapy, and will be indicated by a decrease in skin conductance, an increase in finger temperature, and an increase in heart rate variability. Measurements in the control group will provide a background level of how much physiologic arousal changes with time, independent of music therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hien Duong, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States